CLINICAL TRIAL: NCT01188109
Title: Gemcitabine/Cisplatin for Resected Pancreas Cancer: Establishing the Role of Excision Repair Cross Complementation Gene 1 (ERCC1) in Treatment Decision
Brief Title: Gemcitabine/Cisplatin for Resected Pancreas Cancer: Establishing the Role of ERCC1 in Treatment Decision
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Shishir Kumar Maithel, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00034258; WCI1738-09 (Other: Other)
Record Dates: First submitted 2010-07-23; First posted 2010-08-25 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-08

CONDITIONS: Pancreatic Neoplasms; Pancreatic Cancer
Keywords: Pancreatic Neoplasms; Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine / Cisplatin (Experimental): Single arm study. All patients will receive gemcitabine and cisplatin as adjuvant therapy.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine — Standard of care chemotherapy and dosage
  Dose - 1000 mg/m²
  Schedule - Days 1 and 15; Q 28 days
  Other Names: Gemzar
Drug: Cisplatin — Dose - 50 mg/m²
  Schedule - Days 1 and 15; Q 28 days
  Other Names: Platinol

SUMMARY:
The purpose of this study is to investigate if the investigators can use a specific marker in the pancreatic tumor itself to determine which patients will benefit from receiving combination chemotherapy of gemcitabine and cisplatin after undergoing resection of a pancreatic cancer.

The investigators will also investigate if there is any benefit to receiving both chemotherapy drugs as opposed to only gemcitabine after undergoing complete resection of the tumor.

DETAILED DESCRIPTION:
The study will specifically be looking at ERCC1 expression in pancreas cancer with regards to its prognostic and predictive value as a biomarker for patients receiving Gem / Cis as adjuvant therapy after resection.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 18 years) at the time of signing informed consent form
2. Understand and voluntarily sign informed consent form
3. Able to adhere to study visit schedule and other protocol requirements
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
5. Absolute neutrophil count ≥ 1500 / mm³
6. Platelet count ≥ 100,000 / mm³
7. Resectable pancreatic adenocarcinoma
8. Pathologic diagnosis of pancreatic adenocarcinoma

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing informed consent form
2. A history of renal dysfunction (serum creatinine > 1.8 mg/dL)
3. Presence of active infection
4. Untreated second malignancy
5. Pregnant or breast feeding females (A urine pregnancy test will be obtained in all women of child-bearing age at initial screening prior to study enrollment and administration of chemotherapy.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shishir Maithel, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who underwent resection of a pancreatic adenocarcinoma (PDAC) were enrolled postoperatively at Winship Cancer Institute of Emory University from 2010-2013.
Pre-assignment Details: Twenty-five patients were initially enrolled. Three patients were thereafter excluded; two were diagnosed with secondary malignancies (primary lung adenocarcinoma and thyroid cancer), and one had a diagnosis of cholangiocarcinoma on final surgical pathology.
Groups:
- Gemcitabine / Cisplatin: Single arm study. All patients will receive gemcitabine and cisplatin as adjuvant therapy.
  Gemcitabine: Standard of care chemotherapy and dosage
  Dose - 1000 mg/m²
  Schedule - Days 1 and 15; Q 28 days
  Cisplatin: Dose - 50 mg/m²
  Schedule - Days 1 and 15; Q 28 days
Period: Overall Study
Arm/Group | Gemcitabine / Cisplatin
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine / Cisplatin
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival as Measured by CT Scan
Description: Clinical data were prospectively collected. Staging was performed using 7th American Committee on Cancer criteria. Patients were followed by radiologic evaluation (CT or MRI) and carbohydrate antigen 19-9 (CA19-9) every 3 months for the first 3 years after resection to assess for recurrence. Subsequently, patients underwent imaging every 6 months.
Time Frame: Every 3 months and then every 6 months for 2 more years after resection
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine / Cisplatin
Number analyzed (Participants) | 22
months | 16.7 [6.9 to 26.4]

2. Secondary Outcome: Immunohistochemistry to Determine Status of Excision Repair Cross Complementation Gene-1 (ERCC1) Expression
Description: To determine the level of ERCC1 expression, formalin-fixed, resected tumors were stained with anti-ERCC1 monoclonal antibody (clone 8F1; Neomarkers, Fremont, CA, USA) using the Dako Autostainer (Ft. Collins, CO). The percentage and intensity of fine granular nuclear staining were graded by a single pathologist. Percentage of staining was categorized into the following groups: 0 ≤ 1%; 1 = 1-10%; 2 = 11-50%; 3 = 51-100%. Staining intensity was scored as follows: 0 = none; 1 = weak; 2 = moderate; 3 = strong. Subsequently, an overall score to dichotomize the expression level to low or high was calculated: [(1+intensity score)/3]*percentage score. An overall score ≤ 2 was considered low ERCC1 expression, and > 2 was high ERCC1 expression.
Time Frame: At the time of resection
Population: Twenty patients had tissue available for ERCC1 analysis.
Measure: Number; unit: patients
Arm/Group | Gemcitabine / Cisplatin
Number analyzed (Participants) | 20
patients
  Low Tumor ERCC1 Expression | 15
  High Tumor ERCC1 Expression | 5

ADVERSE EVENTS:
Arm/Group | Gemcitabine / Cisplatin
Serious Adverse Events (participants affected / at risk) | 2/22
Other Adverse Events (participants affected / at risk) | 11/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine / Cisplatin (N=22)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pulmonary Embolus (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine / Cisplatin (N=22)
Fatigue (General disorders) | 1
Nausea/Vomiting (General disorders) | 1
Renal Insufficiency (Renal and urinary disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 8

LIMITATIONS AND CAVEATS:
This study was limited by the small sample size and failure to accrue the 45 patients estimated to appreciate potential differences in outcomes of patients with differential ERCC1 expression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes